CLINICAL TRIAL: NCT06920706
Title: Efficacy of Remote Ischemic Conditioning in Preventing Post-Stroke Depression: A Multicenter, Randomized, Double-Blind, Sham-Controlled Clinical Trial
Brief Title: Efficacy of Remote Ischemic Conditioning in Preventing Post-Stroke Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LYS[2025]039-002
Record Dates: First submitted 2025-03-18; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Post-stroke Depression; Remote Ischemic Conditioning

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- RIC group (Experimental): Subjects in the RIC group receive standard therapy and RIC treatment.
  Interventions: Device: RIC
- Sham-RIC group (Sham Comparator): Subjects in the Sham-RIC group receive standard therapy and Sham-RIC treatment.
  Interventions: Device: Sham-RIC

INTERVENTIONS:
Device: RIC — The ischemic preconditioning training device is applied to the subjects' upper arms to administer pressure (200 mmHg). The pressure is maintained for 5 minutes, followed by 5 minutes of release, completing one ischemia-reperfusion cycle. Each training session consists of 5 consecutive cycles, performed twice daily for 14 days.
  Arms: RIC group
Device: Sham-RIC — The ischemic preconditioning training device is applied to the subjects' upper arms to administer pressure (60 mmHg). The pressure is maintained for 5 minutes, followed by 5 minutes of release, completing one ischemia-reperfusion cycle. Each training session consists of 5 consecutive cycles, performed twice daily for 14 days.
  Arms: Sham-RIC group

SUMMARY:
Post-stroke depression (PSD) is characterized primarily by low mood and loss of interest following a stroke. It is one of the most common and serious complications of stroke, with an incidence of 11% to 41% within two years post-stroke. PSD significantly impacts stroke prognosis, not only hindering neurological recovery but also increasing clinical disability and mortality rates, thereby imposing substantial economic and psychological burdens on families and society. Therefore, preventing PSD is crucial for stroke rehabilitation.

Clinical trials have demonstrated that preventive antidepressant treatment can reduce PSD incidence and improve clinical outcomes; however, controversies remain regarding the timing, methods, and safety. Meanwhile, preventive psychological therapy faces challenges in implementation due to effectiveness, accessibility, and cost-effectiveness.

Remote ischemic preconditioning (RIC) is a non-invasive, cost-effective, and non-pharmacological intervention. By modulating small molecules in the peripheral and central nervous systems through transient, periodic limb blood flow restriction and reperfusion, RIC reverses neurobiological changes and demonstrates neuroprotective potential in various neurological diseases. Recently, a study showed that RIC is safe and effective in preventing PSD; however, the sample size is small and the specific mechanisms remain unclear. Therefore, this study aims to further explore the role and mechanisms of RIC in PSD prevention.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, sham controlled clinical study will enroll acute ischemic stroke patients within 48 hours of symptom onset. Eligible participants will be randomly allocated (1:1) to receive either remote ischemic conditioning (RIC) or sham-RIC treatment for 14 consecutive days. The primary outcome is the incidence of post-stroke depression at day 14 post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient age≥18 years;
* No gender preference;
* Diagnosed with acute ischemic stroke;
* From onset to treatment ≤48 h;
* 6≤ NIHSS scores ≤25;
* Premorbid mRS ≤1;
* Signed informed consent.

Exclusion Criteria:

* Baseline HAMD-24 scores ≥8;
* Infarction area overlapped with the area where the DTI-ALPS index is calculated;
* A history of severe mental illness such as depression, bipolar disorder, and schizophrenia;
* A history of mental disorders caused by other organic diseases, such as post-Parkinson depression;
* Participants with cognitive impairment, disturbance of consciousness, severe hearing impairment, or aphasia who were unable to cooperate with the assessment;
* A history of autoimmune diseases (such as multiple sclerosis, neuromyelitis optica spectrum disorders, systemic lupus erythematosus, etc.), malignant tumors, or obstructive sleep apnea hypopnea syndrome;
* Intracranial tumor, arteriovenous malformation, or aneurysm;
* Uncontrolled severe hypertension (systolic pressure >180mmHg or diastolic pressure >110 mmHg after drug treatment) ;
* Subclavian artery stenosis≥50% or subclavian steal syndrome;
* Any contraindication for remote ischemic adaptation: the upper limb has serious soft tissue injury, fracture or vascular injury, distal upper limb perivascular lesions, etc.;
* Severe coagulation dysfunction, platelet count < 100×10^9/L, cardiac dysfunction (NYHA class Ⅲ or above), hepatic dysfunction (aspartate aminotransferase and/or alanine aminotransferase > 3 times the upper limit of normal), or renal dysfunction (serum creatinine > 265μmol/L);
* Any contraindication for magnetic resonance imaging: metal implants, claustrophobia, etc.;
* Women known to be pregnant or lactating, or have a positive pregnancy test;
* Participating in other clinical trials within three months;
* Participants not suitable for this clinical studies considered by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-stroke depression | Day 14
  The diagnosis of post-stroke depression is established according to the "Depressive Disorder Due to Another Medical Condition" criteria specified in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), using the Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5-RV).

SECONDARY OUTCOMES:
Cumulative incidence of post-stroke depression | Day 28, Day 90, and Day 180
  The cumulative incidence of post-stroke depression is calculated as (number of post-stroke depression cases during follow-up / total enrolled participants) × 100%.
Incidence of post-stroke anxiety | Day 180
  The diagnosis of post-stroke anxiety is established according to the "Anxiety Disorder Due to Another Medical Condition" criteria specified in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), using the Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5-RV).
Cumulative incidence of post-stroke anxiety state | Day 14, Day 28, Day 90, and Day 180
  Post-stroke anxiety state is defined as a 14-item Hamilton Anxiety Rating Scale (HAMA-14) score ≥7 points.
Change from baseline in enlarged perivascular spaces (EPVS) severity score (range 0-4) | Day 14
  EPVS in the basal ganglia (BG) and centrum semiovale (CSO) are visually scored as: 0 = none, 1 = 1-10, 2 = 11-20, 3 = 21-40, and 4 = >40 on the axial slice with the highest burden and hemicerebrum with higher burden. The higher the score, the worse the outcome.
Change from baseline in Diffusion Tensor Imaging-Analysis along the Perivascular Space (DTI-ALPS) index. | Day 14
  The DTI-ALPS index is calculated as the ratio of projection-to-association fiber diffusivity in the lateral ventricular region.
Change from baseline in Neurotransmitter levels in brain regions | Day 14
  Proton magnetic resonance spectroscopy (¹H-MRS) is performed to quantify the levels of N-acetylaspartate (NAA), glutamate/glutamine (Glx), choline (Cho), and creatine (Cr) in the following brain regions: thalamus, caudate nucleus, putamen, globus pallidus, amygdala, hippocampus, insular cortex, medial prefrontal cortex, and cingulate cortex.
Change from baseline in peripheral blood neurotransmitter levels | Day 14
  Levels of γ-aminobutyric acid (GABA), glutamate (Glu), glutamine (Gln), serotonin (5-HT), norepinephrine (NE), and dopamine (DA) in peripheral blood are measured using liquid chromatography-tandem mass spectrometry (LC-MS/MS).
Change from baseline in peripheral blood cytokine levels | Day 14
  Levels of interleukin (IL)-1β, IL-6, IL-10, IL-15, tumor necrosis factor-α (TNF-α), interferon-γ (IFN-γ), and transforming growth factor-β (TGF-β) in peripheral blood are measured using enzyme-linked immunosorbent assay (ELISA).
Change from baseline in 24-item Hamilton Depression Rating Scale (HAMD-24) score (range 0-76) | Day 14, Day 28, Day 90, and Day 180
  The HAMD-24 is a standardized, clinician-rated instrument for quantifying depression severity, where elevated scores correlate with increased symptom burden.
Change from baseline in 14-item Hamilton Anxiety Rating Scale (HAMA-14) score (range 0-56) | Day 14, Day 28, Day 90, and Day 180
  The HAMA-14 is a standardized, clinician-rated instrument for quantifying anxiety severity, with higher scores indicating greater severity.
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) score (range 0-21) | Day 14, Day 28, Day 90, and Day 180
  The PSQI is a validated self-reported questionnaire assessing sleep quality and disturbances over a 1-month period. Higher scores indicate worse sleep quality.
Change from baseline in Fugl-Meyer Assessment (FMA) score (range 0-226) | Day 14
  The FMA is administered to evaluate sensorimotor recovery post-stroke. Higher total scores indicate better functional recovery.
Change from baseline in National Institutes of Health Stroke Scale (NIHSS) score (range 0-42) | Day 14
  The NIHSS is assessed to quantify neurological deficit severity. Higher scores indicate more severe impairment.
Change from baseline in Mini-Mental State Examination (MMSE) score (range 0-30) | Day 90 and Day 180
  The MMSE is administered to assess global cognitive function, with lower scores indicating greater impairment.
Change from baseline in EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) score (range 5-25) | Day 90 and Day 180
  The EQ-5D-5L is administered to assess health-related quality of life. Higher scores indicate worse quality of life.
Change from baseline in EuroQol 5-Dimension 5-Level questionnaire Visual Analogue Scale (EQ-5D-5L VAS) score (range 0-100) | Day 90 and Day 180
  The EQ-5D-5L VAS records self-rated overall health status on a vertical scale, with higher scores indicating better perceived health.
The proportion of modified Rankin Scale (mRS) Score 0-2 | Day 90 and Day 180
  The mRS is administered to evaluate global functional outcomes after stroke, with scores ranging from 0 (no symptoms) to 6 (death). For analysis, outcomes were dichotomized as favorable (mRS 0-2) or poor (mRS 3-6).
The distribution of modified Rankin Scale (mRS) Score (range 0-6) | Day 90 and Day 180
  The mRS is administered to evaluate global functional outcomes after stroke, with higher scores indicating worse outcome.
All-cause mortality | Day 180
  All-cause mortality is defined as death from any cause occurring during the study period.
Total hospitalization time | Day 180
  Total hospitalization time is calculated by summing all inpatient days across neurology and rehabilitation departments within the follow-up period.

OTHER OUTCOMES:
Incidence of adverse events | Day 14, Day 28, Day 90, and Day 180
  Adverse events include dizziness, headache, palpitation, and subcutaneous ecchymosis and swelling at the intervention site.
Incidence of serious adverse events | Day 14, Day 28, Day 90, and Day 180
  Serious adverse events include death, life-threatening illness or injury, hospitalization or prolonged hospitalization, medical or surgical intervention required to prevent permanent injury, severe disability, or incompetence, and other serious medical events.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Jia, Study Director — Xuanwu Hospital, Beijing
Locations (5):
- China (5):
  - Tongren City People's Hospital, Tongren, Guizhou
  - Baoding People's Hospital, Baoding, Hebei
  - Jilin People's Hospital, Jilin, Jilin
  - Jincheng People's Hospital, Jincheng, Shanxi
  - Xuanwu Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No